CLINICAL TRIAL: NCT01222338
Title: Phase 2 Placebo-controlled, Randomized Study of Oral Immunomodulator in TB and TB/HIV Patients
Brief Title: Safety and Efficacy of Oral Immunomodulator in Tuberculosis (TB) and TB/HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisichansk Regional Tuberculosis Dispensary (Other)
Collaborators: National Medical University, Ukraine (Other); Immunitor USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: imm01
Record Dates: First submitted 2010-06-30; First posted 2010-10-18 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Tuberculosis
Keywords: Mycobacterium; MDR-TB; XDR-TB; HIV; HCV
MeSH Terms: conditions — Tuberculosis; Mycobacterium Infections; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis | interventions — V-5 immunitor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunomodulator intervention (Active Comparator): Two cohorts or arms of at least 60 subjects each (total 120) with pulmonary TB positive for sputum AFB smear will be randomized in a 1:1 ratio to receive once-daily, tablet of V-5 immunitor in combination with standard ATT for 2 months followed by ATT outside of trial for next 4 months or however long it needs to be.
  Interventions: Biological: V-5 immunitor
- placebo (Placebo Comparator): Control Cohort 1 (60 subjects) will receive standard first-line ATT regimen: (daily Isoniazide (H) 150mg, Rifampicin (R) 300mg, Ethambutol (E) 400mg, and Pyrazinamide (Z) 400mg during first 2 months, followed by H/R three times per week for the next 4 months. Patients also will receive placebo preparation, appearing identical to V-5 immunitor, taken once daily 30 minutes prior or after meal for 2 months
  Interventions: Biological: V-5 immunitor

INTERVENTIONS:
Biological: V-5 immunitor — once per day dosing for 2 months
  Other Names: V5, V-5 immunitor

SUMMARY:
Treatment of multidrug-resistant TB (MDR-TB) is 100 times more expensive than treatment of drug-susceptible TB, requiring intensive clinical management for prolonged time (18-24 months) and more toxic treatment course. In prior open label study the investigators have shown that adding V-5 Immunitor (V5), can reduce treatment duration to one month and enhance by 4-5 fold the efficacy of TB drugs. Furthermore, V5 has been shown to reverse or reduce liver damage caused by chemotherapy. The cost of V5 will be very modest. The investigators propose to conduct placebo-controlled clinical trial in patients with treatment refractory TB so that the clinical benefit of V5 is confirmed.

DETAILED DESCRIPTION:
The first-diagnosed Mycobacterium tuberculosis infection (TB) is curable with the first line of anti-tuberculosis drugs (ATT) in over 90% of cases within 6 months. The treatment of TB, refractory to conventional ATT, requires the deployment of second line TB drugs. This represents a significant challenge, particularly in resource-poor countries.

The incidence of TB in Ukraine prior to 1992 was about 40 cases per 100,000 people. Ten years later, TB cases increased to over 80/100,000, with mortality doubled from 10.2/100,000 to 21.6/100,000. Drug-resistant TB is now common in Ukraine. Isoniazid and rifampicin resistance, which defines the MDR-TB, has been found in 44% and 32.9% of TB isolates. The first Ukrainian case of HIV was reported in 1987. Today, Ukraine has the highest HIV rate in the Eastern Europe, with increasing proportion of dual infection. For example, in 2002 the prevalence of TB and HIV co-infection was 6.3%, but in 2006 at least 15.5 % of TB patients had HIV co-infection.

It is clear that alternative and improved treatment options are needed. If such an intervention is found, the impact on the healthcare and clinical management of treatment-refractory TB and TB-HIV patients will be tremendous. The significant efforts are directed at finding new drugs and vaccines against TB. Immune-based interventions are actively sought as an adjunct therapy to conventional ATT. In earlier study the investigators have accidentally observed that when patients with chronic hepatitis C and HIV-TB were given V5 together with TB drugs it resulted in negative sputum conversion in 95% of patients within one month. This startling finding had prompted this study. The aim of the present study is to compare the clinical benefit of TB therapy in combination with V5 versus combination of placebo with ATT in a representative population of patients who are poorly manageable due to relapsing TB, MDR-TB, or TB-HIV co-infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years old and are willing and capable of providing written-informed consent.
* Both men and non-pregnant women will be included.
* One group of 30 patients will have HIV.
* Another group of 30 patients will have drug-resistant TB (MDR or XDR).
* Remaining 60 patients will have drug-sensitive TB of which 30 will be assigned to placebo.
* TB infection documented prior to Study Entry by either the presence of TB rapid test or sputum smear positive for acid-fast bacilli (AFB).
* At least two independent tests are sought to confirm TB diagnosis.
* Agreement to participate in the study and to give a sample of blood for HIV testing.

Exclusion Criteria:

* Subjects who have already taken V5 in prior trial and those without baseline data.
* Those who met inclusion criteria can be retrospectively enrolled.
* Those who are re-treated and relapsed will be eligible as long as they are on the same drug regimen as the rest of patients.
* Pregnant or breast-feeding women are excluded.
* Subjects who have taken anti-retroviral drugs or immunomodulatory therapies within 2 months prior to Entry:

  * systemic corticosteroids
  * immune globulin (IV gamma globulin, IVIG)
  * interferons,
  * interleukins
  * pentoxifylline (Trental)
  * thalidomide
  * filgrastim (G-CSF)
  * sargramostim (GM-CSF)
  * dinitrochlorobenzene (DNCB)
  * thymosin alpha 1 (thymosin alpha)
  * thymopentin
  * inosiplex (Isoprinosine)
  * polyribonucleoside (Ampligen)
  * ditiocarb sodium (Imuthiol)
  * any locally available immune modulators
  * and any other therapeutic or preventive vaccine.
* Subjects requiring concurrent participation in another experimental research treatment study, or who received an experimental agent within four weeks prior to Study Entry.
* Medical conditions that in the opinion of the local investigator, may obscure the proper observation of the safety or activity of the study treatment; including any acute medical condition of unknown etiology or recent surgery prior to Entry.
* Medical conditions such as active alcohol or substance abuse, or psychological issues that in the opinion of the local investigator, would interfere with adherence to the requirements of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
primary endpoint: sputum smear conversion | 12 months
  Sputum smear conversion at monthly intervals timepoint Rates of pulmonary healing by chest X-ray at the end of study

SECONDARY OUTCOMES:
liver function | 12 months
  To determine the safety of V5+ATT versus ATT+placebo in TB-infected subjects, Standard parameters, e.g., ALT and bilirubin, liver size will be measured.
quality of life | 12 months
  Measure changes in quality of life by TB score questionnaire
hematology parameters | 12 months
  Measure CBC by standard routine methods
weight gain | 12 months
  Measure changes in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Dmytro Butov, MD, Principal Investigator — Kharkiv National Medical University
Locations (1):
- Lisichansk TB Dispensary, Lisichansk, Luhansk Oblast, Ukraine

REFERENCES:
- [Result] DOI 10.2217/imt.12.59
- [Derived] Batbold U, Butov DO, Kutsyna GA, Damdinpurev N, Grinishina EA, Mijiddorj O, Kovolev ME, Baasanjav K, Butova TS, Sandagdorj M, Batbold O, Tseveendorj A, Chunt E, Zaitzeva SI, Stepanenko HL, Makeeva NI, Mospan IV, Pylypchuk VS, Rowe JL, Nyasulu P, Jirathitikal V, Bain AI, Tarakanovskaya MG, Bourinbaiar AS. Double-blind, placebo-controlled, 1:1 randomized Phase III clinical trial of Immunoxel honey lozenges as an adjunct immunotherapy in 269 patients with pulmonary tuberculosis. Immunotherapy. 2017 Jan;9(1):13-24. doi: 10.2217/imt-2016-0079. Epub 2016 Nov 21. PMID 27868466
- [Derived] Arjanova OV, Prihoda ND, Yurchenko LV, Sokolenko NI, Frolov VM, Tarakanovskaya MG, Batdelger D, Jirathitikal V, Bourinbaiar AS. Adjunct oral immunotherapy in patients with re-treated, multidrug-resistant or HIV-coinfected TB. Immunotherapy. 2011 Feb;3(2):181-91. doi: 10.2217/imt.10.96. Epub 2010 Dec 24. PMID 21182457
- See also: Phase 2 trial of V-5 Immunitor (V5) in patients with chronic hepatitis C co-infected with HIV and Mycobacterium tuberculosis — http://omicsonline.org/2157-7560/2157-7560-1-103.php
- See also: doi: 10.4172/2161-1068.S1-001 Therapeutic Vaccination of Treatment-Failed TB Patients on "Palliative" Support Consisting of Isoniazid and Rifampicin — http://www.omicsonline.org/searchresult.php
- See also: Phase IIb randomized trial of adjunct immunotherapy in patients with first-diagnosed tuberculosis, relapsed and multi-drug-resistant (MDR) TB. — http://www.ncbi.nlm.nih.gov/pubmed/21244690
- See also: Immune approaches in tuberculosis therapy: a brief overview. — http://www.ncbi.nlm.nih.gov/pubmed/22397570